CLINICAL TRIAL: NCT00024843
Title: Family Based Interventions: Preschool Children and Parent
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 988; R01HL065133 (NIH)
Record Dates: First submitted 2001-09-28; First posted 2001-09-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To assess the efficacy of a 2-year family-based weight prevention program in a cohort of overweight preschool children and overweight parent pairs.

DETAILED DESCRIPTION:
BACKGROUND:

The proposal targets a population of individuals of great public health importance who are of high risk for weight gain: pre-school children of overweight parents. Family-based interventions are both theoretically and functionally reasonable approaches for use with these subjects, and the choice to focus on both increased physical activity and healthier food choices in the context of the family's environment is appropriate. The decision to include weight management outcomes on the parent as secondary endpoint is strategically wise and may provide important insights into the process of weight management. A broad array of data is to be collected and strong justification is provided for the inclusion of each.

The study is in response to an initiative issued by the National Institute of Diabetes and Digestive and Kidney Diseases and entitled "Innovative Approaches to the Prevention of Obesity". The resulting grant was later reassigned to the National Heart, Lung, and Blood Institute.

DESIGN NARRATIVE:

Approximately fifty child/parent pairs were recruited and randomized evenly to one of two groups: usual care versus an intervention focused on diet and activity strategies that included weekly group visits (24 weeks), biweekly group visits for parents (12 weeks), monthly group visits for parents (6 months) and quarterly group visits (12 months). Cognitive-behavioral therapy was used to guide interventions, which focussed on empowering a parent as the primary medium by which lifestyle changes were made. Major data collection at baseline, twelve, and 24 months included measures of weight; food and activity records; activity monitor recordings; biopsychosocial profiles; blood lipids, glucose, and insulin; process measures; parenting behavior; and child behavior. The primary study outcome measure was age- and gender-appropriate changes in BMI (expressed as a binomial response). Additional outcomes of particular interest were weight changes in the parent, diet and physical activity levels, parenting skills, and biopsychosocial measures.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachiko St. Jeor — University of Nevada, Las Vegas

REFERENCES:
- [Background] St Jeor ST, Perumean-Chaney S, Sigman-Grant M, Williams C, Foreyt J. Family-based interventions for the treatment of childhood obesity. J Am Diet Assoc. 2002 May;102(5):640-4. doi: 10.1016/s0002-8223(02)90146-x. No abstract available. PMID 12008987